CLINICAL TRIAL: NCT05051150
Title: The Use of Epinephrine Infusion for Prophylaxis Against Maternal Hypotension During Cesarean Delivery: a Randomized Controlled Dose-finding Trial
Brief Title: Epinephrine Infusion for Prophylaxis Against Maternal Hypotension During Caesarean Section
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: tachycardia and arrhythmia in the high doses groups 0.05 and 0.07 necessitate stopping the infusion
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-31-2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Post-spinal Hypotension; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- epinephrine 0.03 mcg (Active Comparator)
  Interventions: Drug: Epinephrin 0.03
- epinephrine 0.05 mcg (Active Comparator)
  Interventions: Drug: Epinephrin 0.05
- epinephrine 0.07 mcg (Active Comparator)
  Interventions: Drug: Epinephrin 0.07

INTERVENTIONS:
Drug: Epinephrin 0.03 — epinephrine infusion rate of 0.03 mcg/kg/min will start from subarachnoid injection of local anesthetic until 5-min after baby delivery
  Arms: epinephrine 0.03 mcg
Drug: Epinephrin 0.05 — epinephrine infusion rate of 0.05 mcg/kg/min will start from subarachnoid injection of local anesthetic until 5-min after baby delivery
  Arms: epinephrine 0.05 mcg
Drug: Epinephrin 0.07 — epinephrine infusion rate of 0.07 mcg/kg/min will start from subarachnoid injection of local anesthetic until 5-min after baby delivery
  Arms: epinephrine 0.07 mcg

SUMMARY:
Maternal hypotension after spinal block is a common complication after subarachnoid block in this population. The incidence of maternal hypotension is nearly 60% when prophylactic vasopressors are not used. Therefore, it is highly recommended to use vasopressors, preferably as continuous infusion, for prophylaxis rather than delaying their use until hypotension occurs.

Phenylephrine (PE) is the recommended drug for prophylaxis against hypotension during cesarean delivery; however, the use of PE is commonly associated with decreased heart rate and probably cardiac output because PE is a pure alpha adrenoreceptor agonist . Introduction of NE in obstetric practice had shown favorable maternal and neonatal outcomes and was associated with higher heart rate and cardiac output compared to PE. However, there is still some mothers who develop bradycardia and diminished cardiac output with the use of NE. The most desired scenario during hemodynamic management of mothers during cesarean delivery would achieve the least possible incidences of maternal hypotension, bradycardia and reactive hypertension. Therefore, it is warranted to reach a vasopressor regimen with the most stable hemodynamic profile.

In the last year, epinephrine was reported for the first time in obstetric practice with acceptable safety on the mother and the fetus. However, there is still lack of data about the most appropriate dose for infusion during cesarean delivery. In this study, we aim to compare three prophylactic infusion rates for epinephrine during cesarean delivery.

DETAILED DESCRIPTION:
Upon arrival to the operating room, the patient will be in supine position with left uterine displacement using a wedge below the right buttock. Routine monitoring will be applied (electrocardiography, pulse oximetry, and non-invasive blood pressure monitor). An 18G-cannula will be inserted, and the patients will receive 10 mg metoclopramide, and 50 mg ranitidine. Baseline heart rate and systolic blood pressure will be recorded as the average of three consecutive readings with 2-minutes interval.

Lactated Ringer's solution will be infused at rate of 15 mL/Kg over 10 minutes as a co-load; spinal anesthesia will be achieved by injecting 10 mg of hyperbaric bupivacaine and 20 mcg fentanyl into the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in supine position with left-lateral tilt and the vasopressor infusion will be started.

To maintain the double-blind scheme, the total dosage of epinephrine (mcg) for patients in each group will be calculated and added to the 50 ml syringe and will be infused at rate of 50 mL/hour. The calculated epinephrine dose will be withdrawn using insulin syringe. The vasopressor infusion will be through the same line as the intravenous fluids using a three-way stopcock. the infusion will be stopped when there is tachycardia (>130% of baseline value) and/or reactive hypertension (systolic blood pressure > 120% of baseline), otherwise the infusion will be stopped 5-mins after the baby delivery.

Block success will be assessed after 5 minutes from intrathecal injection of local anesthetic; and will be confirmed if sensory block level is at T4.

Post-spinal hypotension (defined as systolic blood pressure ≤80% of the baseline reading during the period from intrathecal injection to delivery of the fetus) will be managed by administration of 9 mg of ephedrine Severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading) will be managed by administration IV ephedrine 15 mg.

Reactive hypertension (defined as systolic blood pressure ≥120% from the baseline reading) will be managed by stoppage of the infusion till the next systolic blood pressure reading. The infusion will be then re-started at the half of the initial rate, when systolic blood pressure decreases to be within 20% of the baseline reading.

Intraoperative bradycardia (defined as heart rate less than 55 bpm) will be managed by IV atropine bolus (0.5 mg) will be administered.

Fluid administration will be continued up to a maximum of 1.5 liters. An oxytocin bolus (0.5 IU) will be delivered over five seconds after delivery the infused at a rate of 2.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women
* American society of anesthesiologist I or II,
* scheduled for elective cesarean delivery

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction < 50%, heart block, and arrhythmias),
* hypertensive disorders of pregnancy,
* peripartum bleeding,
* coagulation disorders (patients with INR >1.4 and or platelet count < 80000 /dL)
* any contraindication to regional anesthesia,
* baseline systolic blood pressure (SBP) < 100 mmHg will be excluded from the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
the incidence of post-spinal hypotension | 1 minutes after spinal injection until 5-minutes after the baby delivery
  systolic blood pressure less than 80% of baseline value

SECONDARY OUTCOMES:
the incidence of severe post-spinal hypotension | 1 minutes after spinal injection until 5-minutes after the baby delivery
  systolic blood pressure less than 60% of baseline value
the incidence of reactive hypertension | 1 minutes after spinal injection until 5-minutes after the baby delivery
  systolic blood pressure more than 120% of baseline value
total ephedrine dose | 1 minutes after spinal injection until 5-minutes after the baby delivery
  mg
the incidence of tachycardia | 1 minutes after spinal injection until 5-minutes after the baby delivery
  heart rate >130% of baseline value
the incidence of bradycardia | 1 minutes after spinal injection until 5-minutes after the baby delivery
  heart rate < 55 bpm
number of physician intervention | 1 minutes after spinal injection until 5-minutes after the baby delivery
  stopping or restarting the norepinephrine infusion, or injecting ephedrine or atropine

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt